CLINICAL TRIAL: NCT04947631
Title: A Multi-center, Randomized, Double-blinded, Double-dummy, Parallel Group, 48-week, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DKF-313 in Patients With Benign Prostatic Hyperplasia
Brief Title: Efficacy and Safety of DKF-313 in Patients With Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dongkook Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DKF-313-P3
Record Dates: First submitted 2021-05-19; First posted 2021-07-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tadalafil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DKF-313 (Experimental): Dutasteride 0.5mg + Tadalafil 5mg
  Interventions: Drug: DKF-313; Drug: Dutasteride placebo; Drug: Tadalafil placebo
- Dutasteride (Active Comparator): Dutasteride 0.5mg
  Interventions: Drug: Dutasteride; Drug: DKF-313 placebo; Drug: Tadalafil placebo
- Tadalafil (Active Comparator): Tadalafil 5mg
  Interventions: Drug: Tadalafil; Drug: DKF-313 placebo; Drug: Dutasteride placebo

INTERVENTIONS:
Drug: DKF-313 — Combination of dutasteride 0.5 mg and tadalafil 5 mg once daily for 48 weeks
  Arms: DKF-313
Drug: Dutasteride — Dutasteride 0.5 mg once daily for 48 weeks
  Other Names: Avodart
  Arms: Dutasteride
Drug: Tadalafil — Tadalafil 5 mg once daily for 48 weeks
  Other Names: Cialis
  Arms: Tadalafil
Drug: DKF-313 placebo — Once daily for 48 weeks
  Arms: Dutasteride; Tadalafil
Drug: Dutasteride placebo — Once daily for 48 weeks
  Arms: DKF-313; Tadalafil
Drug: Tadalafil placebo — Once daily for 48 weeks
  Arms: DKF-313; Dutasteride

SUMMARY:
This is a multi-center, randomized, double-blinded, double-dummy, parallel group, 48-week study to evaluated the efficacy and safety of DKF-313 (dutasteride and tadalafil) in patients with benign prostatic hyperplasia.

DETAILED DESCRIPTION:
This study is conducted to access whether DKF-313 once daily for 48 weeks is superior to dutasteride 0.5 mg once daily and tadalafil 5 mg once daily each in improving BPH-LUTS as measured by changes in IPSS total scores.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 45 to 80 years
* BPH diagnosis
* Voluntarily signed the informed consent form
* Willing to participate in the study
* Total IPSS 13 or greater at baseline
* Prostate volume 30 cc or greater by TRUS at baseline
* Qmax 4 to 15 mL/s and minimum voided volume 125 mL or greater at baseline

Exclusion Criteria:

* Serum PSA 4 ng/mL or greater with a positive biopsy result
* Malignant urogenital tumors including prostate cancer, bladder cancer, etc.
* Previous prostatic surgery including TURP, balloon dilatation, thermotherapy and stent replacement or other invasive procedures to treat prostate
* Prostate biopsy within 4 weeks of screening
* Use of alpha-blockers, alpha-agonists, phosphodiesterase type 5 (PDE5) inhibitors, antidiuretics, anticholinergics, cholinergics, antispasmodics, nitrates or herbal preparations affecting prostate within 4 weeks of screening, or 5-alpha reductase inhibitors (5-ARIs) within 24 weeks of screening
* Acute urinary retention within 12 weeks of screening
* Any causes other than BPH resulting in urinary symptoms or changes in flow rate (e.g. neurogenic bladder, bladder neck contracture, urethral stricture, bladder malignancy, acute or chronic prostatitis, acute or chronic urinary tract infections)
* Bladder postvoid residual 200 mL or greater
* Anatomical deformation of the penis (such as angulation, cavernosal fibrosis, or Peyronie's disease) or conditions that might predispose to priapism (such as sickle cell anemia, multiple myeloma, or leukemia)
* Cardiovascular diseases such as myocardial infarction within 12 weeks of screening, unstable angina or angina during sexual intercourse, heart failure (NYHA Class 2 or higher) within 24 weeks of screening, uncontrolled arrhythmias, hypotension (<90/50 mmHg) or uncontrolled hypertension (>170/100 mmHg), or stroke within 24 weeks of screening
* Left ventricular outflow obstruction (e.g. aortic stenosis and idiopathic hypertrophic subaortic stenosis)
* Inherited disorders including galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Inherited retinal degeneration including retinitis pigmentosa
* Vision loss in one eye due to non-arteritic anterior ischemic optic neuropathy (NAION)
* Hypersensitivity to ingredients of investigational products
* Alcohol or drug abuse or treating psychiatric disorders
* Severe hepatic impairment (ALT or AST > 3xULN)
* Renal impairment with severe heart failure (serum creatinine > 2xULN)
* Uncontrolled diabetes (HbA1c 9% or greater)
* Other investigational products or procedures within 12 weeks of screening
* Plans to have a child or unwilling to comply with using medically accepted contraception methods (such as surgical sterilization and condom) during the treatment period
* Not eligible due to other reasons at the investigator's discretion

Ages: 45 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Change in Total International Prostate Symptom Score (IPSS) from baseline to Week 48 | Weeks 0 and 48

SECONDARY OUTCOMES:
Change in Total International Prostate Symptom Score (IPSS) from baseline to Weeks 4, 12, 24 and 36 | Weeks 0, 4, 12, 24 and 36
Change in Total International Prostate Symptom Score (IPSS) voiding (obstructive) subscores from baseline to Weeks 4, 12, 24, 36 and 48 | Weeks 0, 4, 12, 24, 36 and 48
Change in Total International Prostate Symptom Score (IPSS) storage (irritative) subscores from baseline to Weeks 4, 12, 24, 36 and 48 | Weeks 0, 4, 12, 24, 36 and 48
Change in Total International Prostate Symptom Score (IPSS) Quality of Life (QoL) index from baseline to Weeks 4, 12, 24, 36 and 48 | Weeks 0, 4, 12, 24, 36 and 48
Change in Qmax from baseline to Weeks 24 and 48 | Weeks 0, 24 and 48
Change in post void residual (PVR) volume from baseline to Weeks 24 and 48 | Weeks 0, 24 and 48
Change in prostate volume (PV) from baseline to Week 48 | Weeks 0 and 48
Change in prostate specific antigen (PSA) from baseline to Weeks 24 and 48 | Weeks 0, 24 and 48

OTHER OUTCOMES:
Change in International Index of Erectile Function (IIEF) - Erectile Function (EF) domain scores from baseline to Weeks 4, 12, 24, 36 and 48 | Weeks 0, 4, 12, 24, 36 and 48
Change in Sexual Encounter Profile (SEP) Q2 and Q3 from baseline to Weeks 4, 12, 24, 36 and 48 | Weeks 0, 4, 12, 24, 36 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Choung-Soo Kim, M.D.,Ph.D, Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University mokdong Hospital, Seoul, South Korea